CLINICAL TRIAL: NCT07043205
Title: The Psychophysiology of Walking
Acronym: DPVW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Flanders Marine Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0316
Record Dates: First submitted 2025-01-09; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-01

CONDITIONS: Healthy Citizens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 40' walking (Experimental)
  Interventions: Behavioral: Coastal walk; Behavioral: Urban walk

INTERVENTIONS:
Behavioral: Coastal walk — A 40-minute walk with psychophysiological monitoring in Ostend (along the beach)
Behavioral: Urban walk — 40' walk in Ghent (urban)

SUMMARY:
The literature suggests that natural environments, such as those on the Belgian coast, improve several psychological and physiological health parameters. In these environments, recreational activities often involve walking. However, it is still unknown how the effects of the environment and of walking together influence health. This study investigates the effects of a walk on the Belgian coast versus in the city on various psychological and physiological parameters of mental and physical health, both while walking and at rest after walking. A second set of research questions concerns the determination of the mediating roles of the physical activity performed, the other people in the environment, and environmental factors such as weather and perceived safety. This means that the investigators need to measure how these mediators differ between both environments, and to what extent these mediators have an impact on the subjects. A third set of research questions concerns the moderating roles of the individual characteristics (e.g. age, sex, SES personality, health) on the effects.

100 healthy Belgian adult subjects have to take a walk in both environments according to a within-subject cross-over design, while measurements are taken before, during, and after the walks. Before each walk there is also a walking session on a treadmill for baseline measurements, and rest periods before and during the walk to measure responses after the physical activity with the influence of the environment. The walk on the Belgian coast will take place in Ostend on the dike between the beach and the dunes, and the walk in the city will take place in Ghent center on a similar hard surface.

A lot of physiological measurements will be done to determine the activity of the nervous systems and the HPA axis. More specifically, the heart rate will be derived from the electrocardiogram (ECG) as a general measure of the activation of the body and the high-frequency heart rate variability (HF-HRV) as a measure of the change in the activity of the parasympathetic nervous system. From a blood volume pulse signal (BVP) the mean arterial Pressure (MAP) will be derived as a general measure for the activation of the body and the blood circulation. From a skin conductance signal (EDA) the skin conductance level (SCL) and skin conductance responses (SCR) will be derived as measures of the activity of the sympathetic nervous system. From a respiration signal, respiration rate and depth will be derived as measures of regulation by the respiratory center in the brain. The average tone will be derived from the electromyogram (EMG) as a measure of musculoskeletal activation. These electrophysiological measurements will be made using sensors on the body and MindMedia's medically validated Nexus-10 MKII device. The activity of the HPA axis of stress will be measured by determining the concentration of the cortisol hormone in saliva.

In addition, many questionnaires will be administered that measure the stress level, mood, psychological tension (arousal), worrying and rumination, mindfulness-related and subjective experiences of the participants.

The investigators will closely monitor the mediating role of physical activity using a smartphone that will measure accelerometry, location and walking speed. The mediating roles of the other persons in the environment, the weather, and other environmental factors (e.g. naturalness) will be retrospectively questioned via post-walk questionnaires. It is not unimportant that many characteristics of the test subjects can respond to the effect sizes. That is why the investigators also ask for a lot of data about demographics, socio-economic status, lifestyle, health, personality, and other factors for the experiment.

The hypothesis is that as a result of the physical activity, all physiological parameters of stress will increase, because physical activity affects the same physiological pathways as those of stress. The walk on the coast would increase the psychological and physiological differently than the walk in the urban environment. According to the literature, these effects should be are mediated by physical activity, other people in the vicinity, weather, and other environmental factors (e.g. perceived naturalness).

ELIGIBILITY:
Inclusion Criteria:

* speaking dutch
* 18-45 years old
* being a student or having a paid job
* being able to walk for 1 hour

Exclusion Criteria:

* not having a chronic mental or physical condition
* not taking antidepressant drugs
* not being pregnant
* having no uncorrected sensory impairments

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Heart rate in number of beats per minute. | Monitored continuously. Outcome calculated for 2-minute intervals during the different stages of the experiment (i.e., baseline, during walk, during rest after walk; e.g., for two 2-minute intervals during 5-minute baseline).
  Derived from electrocardiogram
High frequency hart rate variability with unit ms² | Monitored continuously. Outcome calculated for 2-minute intervals during the different stages of the experiment (i.e., baseline, during walk, during rest after walk; e.g., for two 2-minute intervals during 5-minute baseline).
  Derived from electrocardiogram
Mean arterial blood pressure in unit µV | Monitored continuously. Outcome calculated for 2-minute intervals during the different stages of the experiment (i.e., baseline, during walk, during rest after walk; e.g., for two 2-minute intervals during 5-minute baseline).
  Derived from blood volume pulse
Skin conductance level in µV | Monitored continuously. Outcome calculated for 2-minute intervals during the different stages of the experiment (i.e., baseline, during walk, during rest after walk; e.g., for two 2-minute intervals during 5-minute baseline).
  Derived from skin conductance signal
Skin conductance response in muS | Monitored continuously. Outcome calculated for 2-minute intervals during the different stages of the experiment (i.e., baseline, during walk, during rest after walk; e.g., for two 2-minute intervals during 5-minute baseline).
  Derived from skin conductance signal
Respiration rate (breaths/minute) | Monitored continuously. Outcome calculated for 2-minute intervals during the different stages of the experiment (i.e., baseline, during walk, during rest after walk; e.g., for two 2-minute intervals during 5-minute baseline).
  Derived from respiration signal
Respiration depth in µV | Monitored continuously. Outcome calculated for 2-minute intervals during the different stages of the experiment (i.e., baseline, during walk, during rest after walk; e.g., for two 2-minute intervals during 5-minute baseline).
  Derived from respiration signal
Average muscle tone in µV | Monitored continuously. Outcome calculated for 2-minute intervals during the different stages of the experiment (i.e., baseline, during walk, during rest after walk; e.g., for two 2-minute intervals during 5-minute baseline).
  Derived from Electromyography
salivary cortisol concentration in nmol/l | Monitored continuously. Outcome calculated for 2-minute intervals during the different stages of the experiment (i.e., baseline, during walk, during rest after walk; e.g., for two 2-minute intervals during 5-minute baseline).
  Derived from saliva
Stress level (1 item VAS 1-10, higher values mean more stress) | Through study completion, an average of 2 hours
  Assessed via questionnaire
Positive mood (10 items, scale 1-5, larger is more positive mood) | Through study completion, an average of 2 hours
  Assessed via questionnaire Positive and Negative Affect Scale (PANAS)
Negative mood (10 items, scale 1-5, larger is more negative mood) | Through study completion, an average of 2 hours
  Assessed via questionnaire Positive and Negative Affect Scale (PANAS)
Arousal level (20 items, scale 1-4, larger is more arousal) | Through study completion, an average of 2 hours
  Assessed via questionnaire Activation-Deactivation Adjective; AD ACL

SECONDARY OUTCOMES:
x, y, z accelerometry in m/s² | Through study completion, an average of 2 hours
  Assessed via accelerometer in smartphone
GPS location in coordinates | Through study completion, an average of 2 hours
  Assessed via GPS in smartphone
Walking speed in m/s | Through study completion, an average of 2 hours
  Assessed via GPS in smartphone

OTHER OUTCOMES:
Perceived naturalness of the environment (VAS, 1-10, higher is more natural) | Through study completion, an average of 2 hours
  Assessed via questionnaire
Enjoyment of weather (VAS, 1-10, higher is more enjoying) | Through study completion, an average of 2 hours
  Assessed via questionnaire
Enjoyment of other people in environment (VAS, 1-10, higher is more enjoying) | Through study completion, an average of 2 hours
  Assessed via questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, East-Flanders, Belgium

REFERENCES:
- See also: Preregistration on OSF — https://osf.io/kzq2e/